CLINICAL TRIAL: NCT01743391
Title: Hysteroscopy Before in Vitro Fertilization - Does it Improve the Outcome?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, Kristine Juul Hare, PhD, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-4-2012-158
Record Dates: First submitted 2012-12-02; First posted 2012-12-06 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Subfertility; Infertility
Keywords: IVF treatment; Office-hysteroscopy; Endometrial biopsy
MeSH Terms: conditions — Infertility | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard treatment
- Intervention (Experimental): Office-hysteroscopy with endometrial biopsy before standard treatment
  Interventions: Procedure: Office-hysteroscopy with biopsy

INTERVENTIONS:
Procedure: Office-hysteroscopy with biopsy
  Arms: Intervention

SUMMARY:
By randomizing sub-fertile women to either control or office-hysteroscopy in the circle prior to IVF or ICSI (intracytoplasmatic sperm injection

) treatment, we aim to enlighten whether hysteroscopy with endometrial biopsy increases pregnancy rates in the intervention group.

DETAILED DESCRIPTION:
Background A tenth of a population in Denmark today is the result of assisted fertility, including IVF and ICSI. In roughly 40 % of these subfertile women the reason is unknown. Standard initial procedures include transvaginal ultrasonography, with or without saline infusion to detect intrauterine abnormalities that might explain the infertile condition. The golden standard to detect intrauterine abnormalities is hysteroscopy. Such abnormalities can be detected in a fourth of this population. Earlier studies indicate that the hysteroscopy alone - without correcting any abnormalities, affects IVF/ISCI outcome positively.

Aim By randomizing patients referred to the fertility clinic to ±office-hysteroscopy in circle prior to IVF/ISCI, we aim to enlighten whether mini-hysteroscopy with endometrial biopsy will increase the fertility by looking at pregnancy rates as our main outcome.

Method Women signed up for second IVF/ISCI treatment will be recruited, after signed consent they are randomized to either office-hysteroscopy or nothing before standard treatment in the fertility clinic.

Mini-hysteroscopy is a standard procedure in our gynecological outpatient clinic. The procedure is done without any anesthetics. Only women with normal intrauterine conditions will be enrolled in this protocol.

When the fertility clinic has a positive serum-HCG (human chorionic gonadotropin

) and a positive transvaginal sonography, pregnancy is confirmed. If negative serum-HCG, negative pregnancy will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Women submitted to IVF or ISCI treatment
* Age > 18 years
* Women able to read, speak and understand Danish
* Written consent

Exclusion Criteria:

* Intrauterine abnormalities
* Infection
* BMI > 35
* Known intrauterine cause to the infertile condition
* Abuse of alcohol or drugs
* Untreated medical condition
* Pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2013-01; Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
pregnancy rates | individual outcome will be evaluated within 8 weeks after IVF treatment. Over all outcome will be evaluated after 3 years.
  Positive serum HCG and transvaginal ultrasonography, alternatively negative serum HCG and negative outcome will be registrated. After 300 women have been included final outcome will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Department of Gynecology and Obstetrics, Copenhagen, Hvidovre, Denmark

REFERENCES:
- [Derived] Berntsen S, Hare KJ, Lossl K, Bogstad J, Palmo J, Praetorius L, Zedeler A, Pinborg A. Endometrial scratch injury with office hysteroscopy before IVF/ICSI: A randomised controlled trial. Eur J Obstet Gynecol Reprod Biol. 2020 Sep;252:112-117. doi: 10.1016/j.ejogrb.2020.06.034. Epub 2020 Jun 17. PMID 32593936